CLINICAL TRIAL: NCT02574416
Title: An Evaluation of the Determinants of Lifestyle and Health Behaviours in Later Life, and to Investigate Their Relationship With Health Outcomes
Brief Title: An Evaluation of the Determinants of Lifestyle and Health Behaviors in Later Life
Acronym: LiLL
Status: Completed | Type: Observational
Sponsor: National Health Service, United Kingdom (Other Government)
Responsible Party: Principal Investigator, Sian Robinson, Professor of Nutritional Epidemiology, National Health Service, United Kingdom
Other Study IDs: RHM MED 1215
Record Dates: First submitted 2015-09-24; First posted 2015-10-12 (Estimated); Last update posted 2018-12-06 (Actual); Status verified 2018-12

CONDITIONS: Aging; Dietary Habits; Life Style
Keywords: Health behaviour; Health outcomes; Diet quality; Physical function; Lifestyle; Older adults
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: There is no intervention — The study is observational and there is no intervention

SUMMARY:
Although increasing age is associated with declining health and function, there are wide variations between individuals in the ageing process. Some of these differences are explained by differences in lifestyle, but little is known about the determinants of lifestyle in older age. The proposed project will describe influences on health behaviour and lifestyle in older adults. Investigators will undertake a prospective study of community-dwelling older people who use any of the Medicine for Older People Services in Southampton, allowing us to gain obtain important insights into the relationship between health behaviour, lifestyle and health outcomes in older people. Our principal aim is to identify key points on the ageing pathway when interventions may be best targeted to promote health. The findings of this project will underpin the design for a complex intervention to be conducted in the future to improve the health outcomes of older people.

DETAILED DESCRIPTION:
Patients will be identified by the Medicine for Older People clinician and asked if they would like to speak to a member of the research team. A member of the research team will approach suitable patients and ask them if they wish to participate. Patients will have the opportunity to read and take away a Patient Information Sheet, and also ask questions about the study and what participating in it would involve. Participants in the study will be telephoned to arrange an appointment for a home visit at a convenient time, or an appointment will be made at this first meeting if this is possible. Written informed consent will be taken at the home visit.

Patients who have used the same Medicine for Older People Services in Southampton within the previous year will be known to the medical team. The medical team will write to the patient with a letter of invitation to participate in the study and the Patient Information Sheet. The letter will contain a reply slip and a stamped addressed envelope. It will also contain contact details should the patient wish to talk to someone about the study and what it would mean for them to participate. Patients who send back their reply slip saying that they would like to participate in the study will be contacted to arrange a home visit at a convenient time. If no reply slip is received after two weeks then a member of the research team will telephone the patient once to find out whether they have received the letter and to offer them the opportunity to participate. This will be done sensitively and carefully and the patients' wishes will be respected at all times. Written informed consent will be taken at the time of the home visit.

All participants will be visited at home by a member of the research team who will interview the participant to obtain background sociodemographic information and a series of short questionnaires will be administered. Each participant will have an assessment of diet quality, appetite and physical function. In addition, weight, grip strength and physical performance will be measured. Participants will be free to decline any part of the questionnaire or assessment.

Two and a half years after this interview the investigators will check on the hospital administration system if the participant's contact details have changed or if they have died since the initial visit. The investigators will then contact the participant by phone (having gained permission to do this at the original assessment visit) to arrange a home visit when diet quality, appetite and physical function will be reassessed. The investigators' experience from the Southampton Mealtime Assistance Study of contacting older study participants by telephone has shown this to be an effective way of ascertaining if the participant is interested in continuing with the study or would prefer not to. The participant will be given the opportunity to refuse a visit with no pressure applied. At the visit the investigators will also ask about the participants' use of the key community services over the past year. The investigators will also ask permission to access the patient's medical records to obtain details of hospital admissions or outpatient appointments in the intervening year.

ELIGIBILITY:
Inclusion Criteria:

* Any person who has attended a Medicine for Older People Service run by Southampton General Hospital between February 2014 and August 2016.

Exclusion Criteria:

* Unable to give informed consent
* acutely unwell

Ages: 60 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Users of the Medicine for Older People Services in Southampton
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Dietary quality | 2.5 years
  Diet quality, which will be assessed by deriving the participants' prudent diet score from the 20-item Food Frequency Questionnaire.

SECONDARY OUTCOMES:
Physical function | 2.5 years
  Physical function which will be assessed by asking ten questions from the Short Form - 36 which ask whether the participants' health limits them from carrying out certain daily activities.
Grip strength | 2.5 years
  Measuring using a Jamar dynamometer
Timed up and go | 2.5 years
  Time taken to rise from a chair, walk 3m and then return to the chair and sit down.
3m walk | 2.5 years
  Time taken to walk 3m
Timed chair rise | 2.5 years
  Time taken to stand up and sit down again five times
Mortality | At 1 year and 2.5 years follow up
  Mortality data will be taken from hospital records
Number of hospital admissions | At one year follow up
  Number of hospital admissions will be abstracted from hospital records
New diagnoses | At one year follow up
  New diagnoses will be taken from hospital records

CONTACTS AND LOCATIONS:
Overall Officials: Sian Robinson, PhD, Principal Investigator — National Health Service, United Kingdom
Locations (1):
- MRC Lifecourse Epidemiology Unit, Southampton, Hampshire, United Kingdom